CLINICAL TRIAL: NCT00118144
Title: Phase II Study of Bortezomib (PS-341) for Patients With Advanced Bronchiolo-Alveolar Carcinoma (BAC) or Adenocarcinoma With BAC Features
Brief Title: Bortezomib in Treating Patients With Stage IIIB or Stage IV Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00113; NCI-2009-00113 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000433404; PHII-57 (Other: City of Hope); 7003 (Other: CTEP); N01CM62208 (NIH); N01CM62201 (NIH); N01CM62209 (NIH); N01CM62207 (NIH)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2013-04

CONDITIONS: Adenocarcinoma of the Lung; Bronchoalveolar Cell Lung Cancer; Non-small Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Bortezomib

ARMS (1):
- Arm I (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1 and 8.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Given IV

SUMMARY:
This phase II trial is studying how well bortezomib works in treating patients with stage IIIB or stage IV lung cancer. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with stage IIIB or IV bronchoalveolar carcinoma (BAC) or adencarcinoma of the lung with BAC features treated with bortezomib.

SECONDARY OBJECTIVES:

I. Determine the progression-free and overall survival of patients treated with this drug.

II. Determine the time to disease progression in patients treated with this drug.

III. Determine predictors of response, based on molecular correlative studies of tumor and blood, in patients with treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to prior epidermal growth factor receptor inhibitor therapy (yes vs no).

Patients receive bortezomib IV over 3-5 seconds on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for survival.

ELIGIBILITY:
Criteria:

* Histologically confirmed bronchoalveolar carcinoma (BAC) or adenocarcinoma of the lung with BAC features:

  * Stage IIIB or IV disease:
  * Patients with stage IIIB disease must be ineligible for definitive combined modality treatment with radiotherapy and chemotherapy
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques or >= 10 mm by spiral CT scan:

  * Previously irradiated lesions are considered measurable only if lesion progressed after completion of radiotherapy
* No unstable brain metastases:

  * Brain metastases that are stable for ≥ 1 month after completion of prior radiotherapy, stereotactic surgery, or surgery are allowed
* Performance status:

  * ECOG 0-2
* Life expectancy >3 months
* Hepatic:

  * Bilirubin normal
  * AST and ALT =< 2.5 times upper limit of normal
* Renal:

  * Creatinine normal OR creatinine clearance >= 60 mL/min
* Cardiovascular:

  * No symptomatic congestive heart failure
  * No unstable angina pectoris
  * No cardiac arrhythmias
* No more than 1 prior chemotherapy regimen for advanced BAC:

  * Prior gefitinib or other known epidermal growth factor receptor (EGFR) inhibitors are not considered a systemic chemotherapy regimen
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* At least 4 weeks since prior corticosteroids
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and for 30 days after completion of study treatment
* No ongoing or active infection
* No other malignancy within the past 3 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer that is in complete remission
* No peripheral neuropathy >= grade 2
* No known hypersensitivity to bortezomib, boron, or mannitol
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No concurrent routine granulocyte colony-stimulating factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])
* At least 2 weeks since prior radiotherapy
* Recovered from prior therapy (alopecia allowed)
* At least 2 weeks since prior EGFR inhibitors
* At least 4 weeks since prior anticonvulsants
* No prior bortezomib
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* Concurrent bisphosphonates for bone metastases allowed
* Hematopoietic:

  * Absolute neutrophil count >= 1,500/mm3
  * Platelet count >= 100,000/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gandara, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients receive bortezomib IV at 1.6 mg/m2 on days 1 and 8 of every 21 day cycle.
Period: Overall Study
Arm/Group | Arm I
Started | 42
Completed | 41
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Patients receive bortezomib IV at 1.6 mg/m2 on days 1 and 8 of every 21 day cycle.
Arm/Group | Arm 1
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 68 [54 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate With Bortezomib Evaluated by Both RECIST Criteria and Computer-assisted Image Analysis.
Description: A response rate of 20% or more with bortezomib would be of interest for further evaluation, whereas a response rate of less than 5% would be of no interest. Response defined as a confirmed CR or PR.
Time Frame: Up to 5 years
Measure: Number; unit: percentage of responders
Arm/Group | Arm 1
Number analyzed (Participants) | 42
percentage of responders | 5

2. Secondary Outcome: Progression-free Survival
Description: Progression Free Survival using the product-limit method of Kaplan and Meier
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1
Number analyzed (Participants) | 42
Months | 5.5 [2.1 to 6.4]

3. Secondary Outcome: Overall Survival
Description: Overall Suvival using the product-limit method of Kaplan and Meier.
Time Frame: Up to 5 years
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Arm I
Number analyzed (Participants) | 42
Months | 13.6 [4.97 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 12/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=42)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Disease progression (General disorders) | 4 (4)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=42)
Hemoglobin decreased (Blood and lymphatic system disorders) | 15 (92)
Lymphangiopathy NOS (Blood and lymphatic system disorders) | 1 (2)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (4)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Endocrine disorder (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (2)
Flashing vision (Eye disorders) | 1 (3)
Vision blurred (Eye disorders) | 3 (9)
Watering eyes (Eye disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (6)
Abdominal pain (Gastrointestinal disorders) | 8 (13)
Constipation (Gastrointestinal disorders) | 14 (42)
Diarrhea (Gastrointestinal disorders) | 20 (51)
Dyspepsia (Gastrointestinal disorders) | 3 (5)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 22 (48)
Stomach pain (Gastrointestinal disorders) | 2 (2)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (4)
Vomiting (Gastrointestinal disorders) | 11 (18)
Chest pain (General disorders) | 7 (16)
Chills (General disorders) | 1 (1)
Death (General disorders) | 3 (3)
Disease progression (General disorders) | 15 (15)
Edema limbs (General disorders) | 4 (5)
Fatigue (General disorders) | 29 (146)
Fever (General disorders) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1)
Ill-defined disorder (General disorders) | 2 (3)
Pain (General disorders) | 6 (7)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (6)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Lip infection (Infections and infestations) | 2 (3)
Otitis externa (Infections and infestations) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 2 (3)
Upper aerodigestive tract infection (Infections and infestations) | 2 (3)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (4)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (12)
Alkaline phosphatase increased (Investigations) | 5 (15)
Aspartate aminotransferase increased (Investigations) | 4 (13)
Bilirubin increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 2 (3)
Hyperbilirubinemia (Investigations) | 1 (3)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (11)
Leukopenia (Investigations) | 3 (25)
Lipase increased (Investigations) | 1 (3)
Lymphocyte count decreased (Investigations) | 9 (9)
Lymphopenia (Investigations) | 3 (7)
Neutrophil count decreased (Investigations) | 6 (28)
Platelet count decreased (Investigations) | 6 (17)
Serum cholesterol increased (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 14 (26)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 10 (28)
Dehydration (Metabolism and nutrition disorders) | 3 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (6)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (11)
Serum albumin decreased (Metabolism and nutrition disorders) | 5 (10)
Serum calcium decreased (Metabolism and nutrition disorders) | 6 (9)
Serum glucose decreased (Metabolism and nutrition disorders) | 3 (3)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (5)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (7)
Serum sodium decreased (Metabolism and nutrition disorders) | 7 (8)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (3)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 12 (30)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (22)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10)
Ataxia (Nervous system disorders) | 1 (5)
Dizziness (Nervous system disorders) | 6 (18)
Headache (Nervous system disorders) | 11 (33)
Memory impairment (Nervous system disorders) | 2 (3)
Neuralgia (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (66)
Seizure (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (3)
Syncope (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (6)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (6)
Insomnia (Psychiatric disorders) | 5 (18)
Protein urine positive (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (16)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (42)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 (51)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (27)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 7 (15)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (4)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 3 (15)
Flushing (Vascular disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (2)
Hot flashes (Vascular disorders) | 1 (6)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less